CLINICAL TRIAL: NCT07049263
Title: Disparities In Access to the Northwest Ambulance Service During Pregnancy, Birth and Postpartum Period and Its Association With Neonatal and Maternal Outcomes [DIAAS]
Brief Title: Disparities In Access to the Northwest Ambulance Service During Pregnancy, Birth and Postpartum Period and Its Association With Neonatal and Maternal Outcomes
Acronym: DIAAS
Status: Active, not recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Stephanie Heys, Chief Investigator and Consultant Midwife (North West Ambulance Service NHS Foundation Trust), Manchester University NHS Foundation Trust
Other Study IDs: G90058; NIHR206378 (Other Grant/Funding Number: NIHR - Research For Patient Benefit (RFPB) Programme)
Record Dates: First submitted 2025-06-20; First posted 2025-07-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Emergency Maternity Care; Health Inequalities in Maternity Care Access; Disparities in Access to Maternity Care; Deprivation; Ethnicity; Ambulances; Pre-hospital
Keywords: Emergency maternity care; Pre-hospital maternity care; Health disparities; Health inequalities; Perinatal period; Maternity care access; Ethnicity; Deprivation; Data linkage; Retrospective cohort study; Mixed methods; Pre-hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NWAS Cohort: A cohort of women who were transferred to Manchester University NHS Foundation Trust during the perinatal period by North West Ambulance Services, between August 2022 and August 2024.
- MFT Cohort: A cohort of women who attended Manchester University NHS Foundation Trust for birth between August 2022 and August 2024, but were not transferred by North West Ambulance Services.

SUMMARY:
This study is the first in the United Kingdom (UK) to look at how women and families from different backgrounds use ambulance services during the 'perinatal period' - through pregnancy, birth, and shortly after having a baby. The researchers want to understand whether all women have the same access to urgent and emergency maternity care, and whether there are differences in health outcomes for mothers and babies who use ambulance services.

The study has two parts (called Work-Packages):

Work Package One will look at data from women who were taken by ambulance to a Manchester University National Health Service (NHS) Foundation Trust (MFT) maternity unit during the perinatal period, compared with those who had a baby at MFT but were not taken there by ambulance. It will look at the differences between the two groups and their health outcomes.

Work Package Two will look closely at the text written by paramedics within ambulance records for some women from Work Package One, especially those at increased risk of a poor outcome. The researchers will study what happened during their care journey and look for anything that happens repeatedly within the text to better understand their experiences.

By combining the results from both work packages, the study aims to give a detailed picture of how different women access emergency maternity care and outcomes for themselves and their babies. This will help identify ways to improve services, especially for women who may face barriers to getting the care they need, helping to make sure that maternity care is safe, fair, and more effective for everyone.

DETAILED DESCRIPTION:
Background:

This study will be the first United Kingdom (UK)-based study to investigate access to ambulance services for women and families from diverse backgrounds during pregnancy, birth and early postpartum period. The study will explore relevant maternal and infant outcomes for families who seek help from the ambulance service to explore health disparities in accessing urgent and emergency care. Findings from this study will inform local and national policy aimed at reducing maternal and perinatal mortality and morbidity. This will contribute to the identification of access challenges experienced by seldom-heard women in a crucially important, but under investigated area of unscheduled urgent and emergency maternity care.

Methods:

A mixed methods approach including two work packages (WP). WP1 includes a retrospective comparative cohort study (WP1) to describe the characteristics of and outcomes for pregnant women and their neonates who are transferred via ambulance to Manchester University National Health Service (NHS) Foundation Trust (MFT) and those that are not. Descriptive statistics with comparative analyses will be presented. WP2 includes a qualitative framework analysis of a purposive sub-sample of routinely collected free-text digital records documented by paramedics for women who arrived at the unit via ambulance. Purposive sampling will be undertaken for women who are identified at an increased risk of poor maternal and/or neonatal outcomes following WP1 analyses. The patient journey will be mapped, and patient profiles constructed. An explanatory mixed methods approach will be undertaken for triangulation of data for insight.

Discussion:

The study aims to provide an in-depth understanding of access to emergency maternity care to allow investigation of opportunities for alternative clinical decision making and review of current service provision. This also helps to identify women with increased risk factors for accessing urgent and emergency care as a gateway to maternity services. This will help to address timely access to the most appropriate services, reducing risk factors for adverse maternity and neonatal outcomes and associated impact upon the emergency services. Findings will be used to inform local and national interventions for at risk populations who access ambulance services during pregnancy, birth, and early postpartum. Findings will also support system conversations around the reasons for seeking help from the ambulance service in the perinatal period and ways to improve access and care provisions for underserved communities.

ELIGIBILITY:
Work Package 1

Inclusion Criteria:

1. North West Ambulance Service (NWAS) Cohort:

   * Had at least one pregnancy start and/or gave birth between 1st August 2022 to 31st August 2024
   * Accessed NWAS service in the perinatal period between 1st August 2022 to 31st August 2024, and were subsequently transferred to an Manchester University NHS Foundation Trust (MFT) maternity unit by ambulance (either to Saint Mary's Oxford Road, Saint Mary's Wythenshawe or Saint Mary's North Manchester sites)
   * Can be linked to the HIVE electronic patient record (EPR) database
   * Has an electronic delivery record on the MFT HIVE database
   * Has not opted out of NHS national data opt-out usage.
2. Comparison Manchester University NHS Foundation Trust (MFT) Cohort:

   * Had at least one pregnancy start and/or gave birth between 1st August 2022 to 31st August 2024
   * Not transferred by ambulance to an MFT maternity unit after contacting NWAS during the perinatal period
   * Attended MFT maternity unit for birth (either Saint Marys Oxford Road, Saint Marys Wythenshawe or Saint Mary's North Manchester Sites) and therefore has an electronic birth record on the MFT HIVE EPR database
   * Has not opted out of NHS national data opt-out usage.

Work Package 1

Exclusion Criteria:

* Opted out of NHS national data usage
* No pregnancy start or end date recorded/imputed
* No birth record on the MFT HIVE EPR database
* Was conveyed by ambulance to a non-MFT maternity unit/site.

Work Package 2

Inclusion Criteria:

* Female
* Had at least one pregnancy and/or gave birth between August 2022 to August 2024
* Accessed NWAS service in the perinatal period between August 2022 to August 2024, and subsequently transferred to an MFT maternity unit by ambulance (either St Marys Oxford Road, St Marys Wythenshawe or North Manchester Sites)
* Has not opted out of NHS national data opt-out usage.

Work Package 2

Exclusion criteria:

- Opted out of NHS national data usage.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Attended a Manchester University NHS Foundation Trust (MFT) maternity unit.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Severe neonatal morbidity (composite) | Up to 6 weeks postpartum.
  Including stillbirth, neonatal death, admission to neonatal intensive care unit, APGAR score <7 at 5 minutes, fetal growth restriction, low arterial cord pH, early preterm birth (<34 weeks), birth injuries and Hypoxic Ischemic Encephalopathy (HIE) diagnosis.
Severe maternal morbidity (composite) | Up to 6 weeks pospartum
  Including maternal death, admission to high dependency or intensive care areas, postnatal hospital readmission, major postpartum haemorrhage (PPH), obstetric anal sphincter injury (OASI), unplanned hysterectomy, placental abruption, eclampsia and Hemolysis Elevated Liver Enzymes and Low Platelets (HELLP) syndrome.

SECONDARY OUTCOMES:
Mode of birth | Up to 6 weeks postpartum.
  Maternal. Spontaneous vaginal birth, breech birth, instrumental birth (forceps, kiwi or ventouse) or Caesarean section birth.
Postpartum Haemorrhage | Up to 6 weeks postpartum
  Maternal. 500ml - 2000ml
Episiotomy | Up to 6 weeks postpartum
  Maternal.
Length of stay in hospital after birth (maternal and neonatal) | Up to 6 weeks postpartum
  Maternal and neonatal. Days.
Number of antenatal visits and ultrasound scans | Up to 6 weeks postpartum
  Maternal.
Need for blood transfusion | Up to 6 weeks postpartum
  Maternal.
Fetal loss <24 weeks' gestation | Up to 6 weeks postpartum
  Maternal.
Maternal death | Up to 6 weeks postpartum
  Maternal.
Admitted to Intensive Care Unit or High Dependency Unit | Up to 6 weeks postpartum
  Maternal. During the perinatal period.
Unplanned hysterectomy | Up to 6 weeks postpartum
  Maternal.
Readmission to hospital in postnatal period | Up to 6 weeks postpartum
  Maternal.
Major Postpartum Haemorrhage | Up to 6 weeks postpartum
  Maternal. >2000mls
Obstetric Anal Sphincter Injury (OASI) | Up to 6 weeks postpartum
  Maternal. Third or fourth degree perineal tear.
Placental abruption | Up to 6 weeks postpartum.
  Maternal.
Eclampsia | Up to 6 weeks postpartum
  Maternal.
Hemolysis, Elevated Liver enzymes and Low Platelets (HELLP syndrome) | Up to 6 weeks postpartum
  Maternal
Stillbirth | Up to 6 weeks postpartum
  Neonatal
Neonatal Death | Up to 28 days after birth.
  Neonatal
APGAR score <7 at 5 minutes | Up to 6 weeks postpartum
  Neonatal
Fetal growth restriction | Up to 6 weeks postpartum
  Neonatal.
Low arterial cord pH at birth | Up to 6 weeks postpartum
  pH <7.05. Neonatal.
Admission to Neonatal Intensive Care Unit (NICU) | Up to 6 weeks postpartum
  Neonatal
Preterm birth | Up to 6 weeks postpartum
  Neonatal. <34 weeks gestation.
Birth-related injury | Up to 6 weeks postpartum
  Neonatal. Including brachial plexus injury, clavicular fractures.
Diagnosis of Hypoxic Ischemic Encephalopathy (HIE) | Up to 6 weeks postpartum
  Neonatal.
Cord prolapse | Up to 6 weeks postpartum
  Maternal
Birth before arrival at hospital (BBA) | Up to 6 weeks postpartum
  Neonatal.
Breastfeeding at discharge | Up to 6 weeks postpartum
  Neonatal.
Low birth weight (LBW) | Up to 6 weeks postpartum
  Neonatal. Grams.
High Birth Weight (HBW) | Up to 6 weeks postpartum
  Neonatal. Grams.
Gestational diabetes | Up to 6 weeks postpartum
  Maternal.
Pre-eclampsia | Up to 6 weeks postpartum
  Maternal.
Antepartum haemorrhage | Up to 6 weeks postpartum.
  Maternal.
Obstetric cholestasis | Up to 6 weeks postpartum
  Maternal.
Venous thromboembolism | Up to 6 weeks postpartum
  Maternal.
Gestational hypertension | Up to 6 weeks postpartum
  Maternal.
Small for Gestational Age (SGA) | Up to 6 weeks postpartum
  Neonatal.
Large for Gestational Age (LGA) | Up to 6 weeks postpartum
  Neonatal.
Low neonatal axillary temperature | Up to 6 weeks postpartum
  Neonatal. On admission. Celcius.
Admitted with COVID-19, RSV, Whooping Cough or Influenza | Up to 6 weeks postpartum.
  Maternal.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be anonymised by the Manchester NHS Foundation Trust (MFT) Clinical Data Science Unit (CDSU) following NHS Data Opt-Out being applied. No personalised patient data will be handled by the DIAAS research team.